CLINICAL TRIAL: NCT05755789
Title: Intermittent Cefoxitin Administration Versus Loading Bolus Followed by Continuous Infusion for the Prevention of Surgical Site Infection in Colorectal Surgery: a Multicentre, Double-blind, Randomized Controlled Clinical Trial
Brief Title: Intermittent Cefoxitin Administration Versus Loading Bolus Followed by Continuous Infusion for the Prevention of Surgical Site Infection in Colorectal Surgery
Acronym: PROPHYLOXITIN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PROPHYLOXITIN
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Antibiotic Prophylaxis; Colorectal Surgery
Keywords: cefoxitin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (innovative administration scheme) (Experimental): Continuous infusion of cefoxitin + Intermittent placebo
  Interventions: Drug: Loading bolus of cefoxitin; Drug: Continuous infusion of cefoxitin; Drug: Intermittent placebo
- Control group (recommended administration scheme) (Active Comparator): Intermittent cefoxitin + Continuous infusion of placebo
  Interventions: Drug: Loading bolus of cefoxitin; Drug: Intermittent cefoxitin; Drug: Continuous infusion of placebo

INTERVENTIONS:
Drug: Loading bolus of cefoxitin — Cefoxitin [2g] before incision
Drug: Intermittent cefoxitin — Additional bolus of cefoxitin [1g] every 2 hours until the end of surgical closure
  Arms: Control group (recommended administration scheme)
Drug: Continuous infusion of placebo — Continuous infusion of placebo from the end of the loading bolus until the end of surgical closure
  Arms: Control group (recommended administration scheme)
Drug: Continuous infusion of cefoxitin — Continuous infusion of cefoxitin [0.5g/h] from the end of the loading bolus until the end of surgical closure
  Arms: Intervention group (innovative administration scheme)
Drug: Intermittent placebo — Additional bolus of placebo every 2 hours until the end of surgical closure
  Arms: Intervention group (innovative administration scheme)

SUMMARY:
The goal of this prospective, multicentre, double-blind, randomized clinical trial is to compare intermittent cefoxitin administration to loading bolus followed by continuous infusion for surgical antibiotic prophylaxis in colorectal surgery.

The main objective is to demonstrate the superiority of a loading dose of cefoxitin followed by continuous infusion over standard of care boluses in reducing SSI within 30 days after colorectal surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Undergoing colorectal surgery (predictable duration > 90 min)

Exclusion Criteria:

* Patients with known history of hypersensitivity to cefoxitin or others beta-lactams
* Patients with extreme severe obesity (defined by a body mass index greater than 50 kg/m2)
* Patients with severe renal insufficiency (clearance creatinine < 30ml/min)
* Active bacterial infection at the time of surgery or recent antimicrobial therapy (up to 2 weeks before surgery) except for oral surgical antibiotic prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | within 30 days after surgery
  Proportion of patients with any surgical site infection according to the CDC criteria

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - Centre Hospitalier de Poitiers, Poitiers, Vienne
  - CHU Angers, Angers
  - Hopital privé Arras les Bonnettes, Arras
  - CHU Caen, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - Centre Léon Bérard, Lyon
  - Hospices Civils Lyon, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHRU Nancy, Nancy
  - CHU de Nantes, Nantes
  - Hopital Européen Gorges Pompidou, Paris
  - Clinique Mutualiste la Sagesse, Rennes
  - Hôpital Privé Rennais Cesson Sevigné, Rennes
  - CH St Brieuc, Saint-Brieuc
  - CHU St Etienne, Saint-Etienne
  - Hopitaux de Strasbourg, Strasbourg
  - CHU Toulouse Rangueil, Toulouse
  - CH Bretagne Atlantique vannes, Vannes

REFERENCES:
- [Derived] Saint-Genis Q, Birckener J, Gourdou V, Nicolle C, Garnier M, Schwindenhammer V, Hannezo C, Aveline C, Cinotti R, Puisney B, Garot M, Chevalier S, Aubert JS, Wodey M, Lasocki S, Lecoeur S, Lagarrigue CJ, Li A, Faucher M, Foucher Y, Frasca D, Boisson M. Multicentre, double-blind, randomised controlled clinical trial comparing intermittent cefoxitin administration versus loading bolus followed by continuous infusion for the prevention of surgical site infection in colorectal surgery: the PROPHYLOXITIN study protocol. BMJ Open. 2025 Jan 28;15(1):e088306. doi: 10.1136/bmjopen-2024-088306. PMID 39880423